CLINICAL TRIAL: NCT07189624
Title: Effect of Acute Endurance Exercise on the Production of FGF21 and Follistatin in Patients With Hepatocellular Carcinoma
Acronym: ECHEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2024 ABERGEL
Record Dates: First submitted 2025-05-16; First posted 2025-09-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis With Hepatocellular Carcinoma
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): A single study visit will be required, during which the following will be caried out:
  * an assessment of physical condition: lower limb isometric strength test, liver frailty index, short physical performance battery, ultrasound assessment of quadriceps muscle mass
  * a 30-minutes exercise session on a bicycle (with heart rate monitor and gas exchange analyzer)
  * 3 fasting blood tests (before, at the end and 1 hour after the exercise) to assess the production of hepatokines and metabolites
  * measurements of perceived fatigue, muscle pain and effort (before, at the end and 1 hour after the exercise).
  Snacks will be served afterwards.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 30-minutes exercise on a bicycle with heart rate monitor and gas exchange analyzer.

SUMMARY:
The main purpose of the study is to characterize the production of hepatokines (FGF21 and Follistatin) in response to a submaximal exercise on an ergocycle, in patients with hepatocellular carcinoma. The effect of exercise on hepatokines and metabolites production in liver cancer patients is not known. Studying this production could help to provide relevant recommendations for training programming in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma developed on cirrhosis
* Cirrhosis of any etiology, defined by a liver elasticity measurement >15kPa or a history of cirrhosis decompensation
* Hepatocellular carcinoma with indication for treatment by immunotherapy or chemoembolization
* Child-Pugh scores A and B7
* WHO score ≤ 2
* Affiliation to french national social security system

Exclusion Criteria:

* Hepatic encephalopathy grade II or higher
* Bone metastasis
* Surgery performed within 30 days prior to inclusion visit
* Liver transplant
* Muscle injury within 3 months of inclusion
* Pregnant or breast-feeding women
* Patients under legal protection (guardianship, curatorship, safeguard of justice)
* Participation in another clinical trial within 10 days of inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Systemic hepatokines rates (FGF-21 and follistatin) | Baseline (pre-exercise), immediately after exercise, 1 hour after the end of exercise
  Blood samples

SECONDARY OUTCOMES:
Muscle pain assessment | Baseline (pre-exercise), immediately after exercise, 1 hour after the end of exercise
  Visual analog scale. Score from 0 (total absence of muscle pain) to 10 (maximum muscle pain).

OTHER OUTCOMES:
Fatigue assessment | Baseline (pre-exercise), immediately after exercise, 1 hour after the end of exercise
  Visual analog scale. Score from 0 (total absence of fatigue) to 10 (maximum fatigue).
Perception of effort assessment | Baseline (at the beginning), periprocedural (middle of exercise), immediately after exercise
  Borg scale
Production of metabolites | Baseline (pre-exercise), immediately after exercise, 1 hour after the end of exercise
  Blood samples

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Estaing Medecine Digestive Et Hepatobiliaire, Clermont-Ferrand
  - CHU de Clermont-Ferrand, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: No